CLINICAL TRIAL: NCT01271634
Title: Observation of the Abnormal Potential From the Offending Vessel to the Facial Muscles of Hemifacial Spasm Patients
Brief Title: Observe Abnormal Potential From the Offending Vessel to the Facial Muscles of HFS Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Xuesheng Zheng, XinHua Hospital, Affiliated to Shanghai JiaoTong University School of Medicine
Other Study IDs: xzheng-hfs-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Hemifacial Spasm
Keywords: cross-transmission; offending vessel
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pathophysiologic basis of hemifacial spasm is cross-transmission between different branches of the facial nerve. The hypothesis is that the cross-transmission is mediated by the sympathetic nerve fibers on the surface of the offending artery. The abnormal potential from the offending vessel to the facial muscles will be detected on hemifacial spasm patients, so as to determine if the sympathetic nerve fibers take part in the circuit of cross-transmission.

DETAILED DESCRIPTION:
It's hypothesized that at the location where the facial nerve is compressed by an artery, ephaptic cross-transmission takes place between the nude facial nerve fibers and the sympathetic nerve fibers on the arterial surface. Thus action potentials could spread indirectly from one facial nerve fiber to several other facial nerve fibers (via the "bridge" of sympathetic fibers), or directly from the sympathetic fibers to facial nerve fibers. The investigators assume this is the electrophysiological basis of hemifacial spasm and its characteristic sign abnormal muscle response (AMR). If an abnormal potential from the offending artery to the facial muscles similar to AMR can be recorded, the hypothesis will be verified.

ELIGIBILITY:
Inclusion Criteria:

1. the age of 18-65 years old;
2. with typical hemifacial spasm symptoms;
3. with typical abnormal muscle response;
4. preoperative magnetic resonance imaging revealed obvious paraneural artery;
5. with informed consent.

Exclusion Criteria:

1. pregnant or lactating women;
2. accompanied by other serious diseases, including liver, kidney, cardiovascular diseases;
3. accompanied by mental illness or severe neurosis;
4. unable to express the subjective symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 20 cases of hemifacial spasm patients who want to undergo microvascular decompression.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Abnormal Potential From the Offending Vessel to the Facial Muscles | up to 4 months

SECONDARY OUTCOMES:
Latency from the root entry zone of facial nerve to the facial muscles | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Xuesheng Zheng, M.D., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- XinHua Hospital, Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Moller AR, Jannetta PJ. On the origin of synkinesis in hemifacial spasm: results of intracranial recordings. J Neurosurg. 1984 Sep;61(3):569-76. doi: 10.3171/jns.1984.61.3.0569. PMID 6086858